CLINICAL TRIAL: NCT04308395
Title: A Phase 3, Multicenter, Open-Label Extension Study of Patidegib Topical Gel, 2% in Subjects With Gorlin Syndrome (Basal Cell Nevus Syndrome)
Brief Title: Extension Study of Patidegib Topical Gel, 2% in Subjects With Gorlin Syndrome (Basal Cell Nevus Syndrome)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated early due to low blinded event rate and this study termination is not related to safety of the drug Patidegib Topical Gel, 2%.
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pelle-926-301E
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-07

CONDITIONS: Basal Cell Nevus Syndrome
Keywords: Gorlin syndrome; Patidegib; Basal cell nevus syndrome; Nevoid basal cell carcinoma syndrome; Basal cell carcinoma; Hedgehog; Surgically eligible basal cell carcinomas; BCC; BCNS
MeSH Terms: conditions — Basal Cell Nevus Syndrome; Carcinoma, Basal Cell

STUDY DESIGN:
Intervention Model Description: All patients will receive Patidegib Topical Gel, 2%,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patidegib Topical Gel, 2% (Experimental): Patidegib Topical Gel, 2%
  Interventions: Drug: Patidegib Topical Gel, 2%

INTERVENTIONS:
Drug: Patidegib Topical Gel, 2% — Patidegib Topical Gel, 2%

SUMMARY:
This is a multicenter, open label extension study evaluating the safety of Patidegib Topical Gel, 2%, applied topically twice daily to the face of adult subjects with Gorlin syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have completed PellePharm Study Pelle-926-201 or Pelle-926-301.
2. Study Pelle-926-301 subjects must have completed the End of Treatment Visit in Study 301, prior to the Screening Visit in this study. They must also complete all Study 301 related procedures prior to the Baseline Visit of this study.
3. The subject must be willing to abstain from application of a non-study topical medication (prescription or over the counter) to facial skin for the duration of the trial except as prescribed by the Investigator. Moisturizers and emollients are allowed. Subjects will be encouraged to use their preferred sunscreen with a sunscreen protection factor (SPF) of at least 30 daily on all exposed skin sites.
4. Female subjects must have a negative pregnancy test. For Study 301 subjects a negative serum pregnancy test result from Study 301 is acceptable if the test was done within 7 days of the Screening Visit of this study.
5. If the subject is a woman of child bearing potential (WOCBP), she must be willing to use birth control methods which may be considered highly effective. Hormonal contraception must be supplemented with a barrier method (preferably condom). Birth control must start prior to Baseline, continue through the duration of the study, and for 30 days after last application of investigational product (IP).
6. If the subject is a male with a female sex partner who is a WOCBP, the subject must be willing to use condoms, even after a vasectomy, starting prior to Baseline, through the duration of the study, and for at least 3 months after the last application of IP.
7. The subject is willing for all facial BCCs to be evaluated and follow treatment recommendations made only by the Investigator.
8. The subject is willing to forego treatment of facial BCCs with anything other than the study IP except when the Investigator believes that delay of treatment of a BCC potentially might compromise the health of the subject. In such instances, the only other allowed form of treatment is surgical.

Exclusion Criteria:

1. The subject has used topical treatment to the face or systemic therapies that might interfere with the evaluation of the study IP.
2. The subject has current, recent (within five half lives of the experimental drug or if half life not known, within the past 6 months prior to the Screening Visit), or planned (while enrolled in this study) participation in an experimental drug study (excluding Study 301).
3. The subject is a WOCBP who is unwilling or unable to comply with pregnancy prevention measures.
4. The subject is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director VP, Clinical Operations, Study Director — PellePharm, Inc.
Locations (36):
- United States (17):
  - PellePharm Investigative Site, Fremont, California
  - PellePharm Investigative Site, Newport Beach, California
  - Yale University, New Haven, Connecticut
  - Pellepharm Investigative Site, Miami, Florida
  - PellePharm Investigative Site, Ormond Beach, Florida
  - PellePharm Investigative Site, Chicago, Illinois
  - Laser & Skin Surgery Center of Indiana, Indianapolis, Indiana
  - Pellepharm Investigative Site, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Midvalley Dermatology, Murray, Utah
- PellePhram Investigative Site, Leuven, Belgium
- PellePharm Investigative Site, Copenhagen, Denmark
- France (3):
  - PellePharm Investigative Site, Lille
  - PellePharm Investigative Site, Nantes
  - Hopital Saint Louis, Paris
- Germany (3):
  - PellePharm Investigative Site, Berlin
  - PellePharm Investigative Site, Munich
  - PellePharm Investigative Site, Münster
- Italy (3):
  - AOU Luigi Vanvitelli, Napoli
  - PellePharm Investigative Site, Rozzano
  - PellePharm Investigative Site, Vicenza
- PellePharm Investigative Site, Maastricht, Netherlands
- Spain (3):
  - PellePharm Investigative Site, Barcelona
  - PellePharm Investigative Site, Madrid
  - PellePharm Investigative Site, Seville
- United Kingdom (4):
  - PellePharm Investigative Site, Glasgow
  - PellePharm Investigative Site, London
  - PellePharm Investigative Site, Manchester
  - PellePharm Investigative Site, Oxford

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patidegib Topical Gel, 2%
Started | 108
Completed | 3
Not Completed | 105

BASELINE CHARACTERISTICS:
Groups:
- Patidegib Topical Gel, 2%,: All study subjects were treated with Patidegib Topical Gel 2% (the investigational medicinal product [IMP]), applied topically twice daily to the face.
Arm/Group | Patidegib Topical Gel, 2%,
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 84
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 8
  Black or African American | 0
  White | 87
  More than one race | 2
  Unknown or Not Reported | 8
Height [Mean (Standard Deviation); unit: cm] — Population: 2 participants missing
  cm
    number analyzed (Participants) | 103
    (all) | 175.9 (10.0)
Weight [Mean (Standard Deviation); unit: kg] | 93.1 (21.4)
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: 2 participants missing
  kg/m2
    number analyzed (Participants) | 103
    (all) | 29.9 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs)
Description: IMP=Investigational medicinal product; Unique adverse event = adverse event of a certain preferred term, counted only once within each subject.
  Related adverse event = adverse event with relationship as Definitely, Probably or Possibly.
Time Frame: 12 months
Measure: Number; unit: Number of subjects
Arm/Group | Patidegib Topical Gel, 2%
Number analyzed (Participants) | 105
Number of subjects
  Number of subjects with at least one adverse event | 46
  Number of subjects with at least one adverse event related to IMP | 6
  Number of subjects with at least leading to treatment discontinuation | 0
  Number of subjects with at least one AE related to IMP leading to treatment discontinuation | 0
  Number of subjects with at least one paralesional adverse event | 3
  Number of subjects with at least one serious adverse event | 3
  Number of subjects with at least one serious adverse event related to IMP | 0
  Number of subjects withat least one adverse event leading to death | 0
  Number of subjects with at least one adverse event related to IMP leading to death | 0

2. Secondary Outcome: Change in Number of Facial BCCs Removed by Surgery
Time Frame: 12 months
Population: Due to the Sponsor's decision to discontinue the trial, no secondary outcomes data was collected
Arm/Group | Patidegib Topical Gel, 2%
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Number of New Lesions Suspicious for BCC
Time Frame: 12 months
Population: Due to the Sponsor's decision to discontinue the trial, no secondary outcomes data was collected
Arm/Group | Patidegib Topical Gel, 2%
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Advanced Basal Cell Carcinoma Index (aBCCdex) Lesion Score
Time Frame: 12 months
Population: Due to the Sponsor's decision to discontinue the trial, no secondary outcomes data was collected
Arm/Group | Patidegib Topical Gel, 2%
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI)
Time Frame: 12 months
Population: Due to the Sponsor's decision to discontinue the trial, no secondary outcomes data was collected
Arm/Group | Patidegib Topical Gel, 2%
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in EuroQol Group 5-level EQ 5D (EQ 5D 5L)
Time Frame: 12 months
Population: Due to the Sponsor's decision to discontinue the trial, no secondary outcomes data was collected
Arm/Group | Patidegib Topical Gel, 2%
Number analyzed (Participants) | 0

7. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs)
Description: as for outcome 1
Time Frame: 12 months
Measure: Number; unit: Number of adverse events
Arm/Group | Patidegib Topical Gel, 2%
Number analyzed (Participants) | 105
Number of adverse events
  Total number of adverse events | 82
  Number of unique adverse events | 72

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Patidegib Topical Gel, 2%
All-Cause Mortality (participants affected / at risk) | 0/105
Serious Adverse Events (participants affected / at risk) | 3/105
Other Adverse Events (participants affected / at risk) | 46/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patidegib Topical Gel, 2% (N=105)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patidegib Topical Gel, 2% (N=105)
No adverse event occured in 5% or more of the patients (General disorders) | 46 (82) — No adverse event occured in 5% or more of the patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT04308395/Prot_002.pdf
  • Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT04308395/SAP_003.pdf